CLINICAL TRIAL: NCT01157091
Title: A Phase II Study of Pazopanib in VEGF-TKI Refractory Metastatic Renal Cell Carcinoma (MRCC)
Brief Title: Pazopanib Hydrochloride in Treating Patients With Stage IV Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10030; NCI-2010-01497
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis; Other: immunologic technique

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given orally
  Other Names: GW786034; Votrient
Other: laboratory biomarker analysis — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological

SUMMARY:
RATIONALE: Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well pazopanib hydrochloride works in treating patients with stage IV kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (RR) associated with pazopanib (pazopanib hydrochloride) as 3rd-line therapy in metastatic renal cell carcinoma (mRCC) patients who have failed therapy with a distinct vascular endothelial growth factor (VEGF)-tyrosine kinase inhibitor (TKI).

SECONDARY OBJECTIVES:

I. To determine if baseline hepatocyte growth factor (HGF), endothelial selectin (E-selectin) and interleukin-6 (IL-6) are associated with progression-free survival (PFS).

II. To determine if pre-metastatic niche density in regional lymph nodes (LNs) is associated with PFS.

III. To determine an association between E-selectin, IL-6 and pre-metastatic niche density.

IV. To evaluate the prognostic effect of pre-metastatic niches as an independent factor in time to first relapse.

V. To determine if phosphorylated signal transducer and activator of transcription 3 (pSTAT3) in tumor tissue is associated with PFS.

VI. To describe the toxicity associated with pazopanib in this patient population.

VII. To evaluate PFS and overall survival (OS). VIII. To compare, within patient, time to tumor progression of 2nd-line therapy with time to tumor progression on pazopanib as 3rd-line therapy.

OUTLINE:

Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion

* Histologically confirmed diagnosis of metastatic clear cell RCC
* At least one measurable lesion at baseline as per RECIST 1.1 criteria; if skin lesions are reported as target lesions, they must be documented (at baseline and at every physical exam) using color photography and a measuring device (such as a caliper) in clear focus to allow the size of the lesion to be determined from the photograph
* 1 prior VEGF-TKI required
* 1 other prior systemic therapy allowed
* ECOG PS 0-1
* Resolution of grade >= 2 toxicity from prior therapy
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* A female is eligible to enter and participate in this study if she is of non-child bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had (1) a hysterectomy, (2) a bilateral oophorectomy (ovariectomy), (3) a bilateral tubal ligation, or (4) is post-menopausal; subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40pg/mL (< 140 pmol/L); subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
* Patients with childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception; GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows: (1) complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product, (2) oral contraceptive, either combined or progestogen alone, (3) injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year, (4) male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject, (6) double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository); female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin >= 9 g/dL (5.6 mmol/L)
* Platelets >= 100 X 10^9/L
* Prothrombin time (PT) or international normalized ratio (INR) =< 1.2 X ULN
* Activated partial thromboplastin time (aPTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN
* Alanine amino transferase (ALT) =< 2.5 X ULN
* Aspartate aminotransferase (AST) =< 2.5 X ULN
* Serum creatinine =< 2.0 mg/dL (133 umol/L) or, if >2.0 mg/dL; calculated creatinine clearance (ClCR) by Cockroft-Gault formula >= 30 mL/min
* Urine Protein to Creatinine Ratio (UPC) < 1

Exclusion

* Concurrent use of other investigational agents
* Known history of allergic reactions to pazopanib or other VEGF-TKIs
* Presence of serious or uncontrolled infection
* Prior malignancy (Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible)
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug; screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to (1) active peptic ulcer disease, (2) known intraluminal metastatic lesion/s with risk of bleeding, (3) inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), (4) other gastrointestinal conditions with increased risk of perforation, or (5) history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to (1) malabsorption syndrome or (2) major resection of the stomach or small bowel
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months: (1) cardiac angioplasty or stenting, (2) myocardial infarction, (3) unstable angina, (4) coronary artery bypass graft surgery, (5) symptomatic peripheral vascular disease, or (6) Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension defined as systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure (DBP) of >= 90mmHg
* Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be < 140/90 mmHg in order for a subject to be eligible for the study
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months; (Note: subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible)
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks prior to the first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications list as specified in the full protocol for at least 14 days of a drug prior to the first dose of study drug and for the duration of the study
* Treatment with any of the following anti-cancer therapies: (1) radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR (2) chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity, except alopecia
* Non-Compliance: Patients, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Medications that inhibit CYP3A4 may result in increased plasma pazopanib concentrations; therefore, co-administration of strong CYP3A4 inhibitors is PROHIBITED beginning 14 days prior to the first dose of study drug until discontinuation from the study; strong CYP3A4 inhibitors include (but are not limited to): certain antibiotics (including clarithromycin, telithromycin, and troleandomycin), certain HIV protease inhibitors (including ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, and lopinavir), certain antifungals (including itraconazole, ketoconazole, voriconazole, and fluconazole) and certain antidepressants (including nefazodone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2013-10-17 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta Pal, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Pazopanib HCl: Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  pazopanib hydrochloride: Given orally
  laboratory biomarker analysis: Correlative studies
  immunologic technique: Correlative studies
Period: Overall Study
Arm/Group | Oral Pazopanib HCl
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 63.1 [45.4 to 86.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Non-Hispanic | 4
  White/Hispanic or Latino | 8
  White/Non-Hispanic | 16
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Complete Response and Partial Response) as Assessed by RECIST 1.1 Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Overall Response (OR) = CR + PR.
Time Frame: 1 year post treatment
Population: Participants with evaluable results.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 25
Participants
  Complete or Partial Response | 14
  Stable | 7
  Progression | 4

2. Secondary Outcome: Progression-free Survival
Description: Kaplan-meier estimate of Progression-free survival, one-year post enrollment in the study. 95% Confidence Intervals are constructed using the Greenwood estimate of variance and log-log transformation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or an unequivocal measured increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year post treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 28
percentage of participants | 70.0 [48.7 to 83.8]

3. Secondary Outcome: Overall Survival
Description: One-year Kaplan-Meier estimate of survival, given in percent, with a 95% Confidence Interval based on the Greenwood variance, with log-log transform.
Time Frame: 1 year post treatment
Population: Patients eligible and enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 28
percentage of participants | 96.0 [72.9 to 99.4]

ADVERSE EVENTS:
Time Frame: 28-day time spans for each cycle. Cycles follow each other until the patient is off-study, up to one year.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 5/28
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=28)
10000081-Abdominal pain (Gastrointestinal disorders) | 1 (1)
10028813-Nausea (Gastrointestinal disorders) | 1 (1)
10016256-Fatigue (General disorders) | 1 (1)
10062501-Non-cardiac chest pain (General disorders) | 1 (1)
10023424-Kidney infection (Infections and infestations) | 1 (1)
10040872-Skin infection (Infections and infestations) | 1 (1)
10046571-Urinary tract infection (Infections and infestations) | 1 (1)
10001675-Alkaline phosphatase increased (Investigations) | 1 (1)
10011368-Creatinine increased (Investigations) | 1 (1)
10025256-Lymphocyte count decreased (Investigations) | 1 (1)
10029366-Neutrophil count decreased (Investigations) | 2 (2)
10035528-Platelet count decreased (Investigations) | 1 (1)
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
10069339-Acute kidney injury (Renal and urinary disorders) | 1 (1)
10020772-Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=28)
10002272-Anemia (Blood and lymphatic system disorders) | 11 (11)
10033557-Palpitations (Cardiac disorders) | 1 (1)
10034474-Pericardial effusion (Cardiac disorders) | 1 (1)
10040741-Sinus bradycardia (Cardiac disorders) | 4 (4)
10040752-Sinus tachycardia (Cardiac disorders) | 7 (7)
aortic sclerosis w/o significant stenosis, mitral annular calcification (Cardiac disorders) | 1 (1)
10005886-Blurred vision (Eye disorders) | 1 (1)
10000081-Abdominal pain (Gastrointestinal disorders) | 7 (7)
10002167-Anal pain (Gastrointestinal disorders) | 1 (1)
10005265-Bloating (Gastrointestinal disorders) | 1 (1)
10009887-Colitis (Gastrointestinal disorders) | 1 (1)
10010774-Constipation (Gastrointestinal disorders) | 6 (6)
10012727-Diarrhea (Gastrointestinal disorders) | 16 (16)
10013781-Dry mouth (Gastrointestinal disorders) | 1 (1)
10016766-Flatulence (Gastrointestinal disorders) | 4 (4)
10017853-Gastritis (Gastrointestinal disorders) | 2 (2)
10019611-Hemorrhoids (Gastrointestinal disorders) | 2 (2)
10028130-Mucositis oral (Gastrointestinal disorders) | 1 (1)
10028813-Nausea (Gastrointestinal disorders) | 14 (14)
10031009-Oral pain (Gastrointestinal disorders) | 1 (1)
10038062-Rectal fistula (Gastrointestinal disorders) | 1 (1)
10038064-Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
10038072-Rectal pain (Gastrointestinal disorders) | 2 (2)
10042112-Stomach pain (Gastrointestinal disorders) | 1 (1)
10047700-Vomiting (Gastrointestinal disorders) | 6 (6)
10054520-Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
10066874-Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
10008531-Chills (General disorders) | 2 (2)
10016256-Fatigue (General disorders) | 16 (16)
10016558-Fever (General disorders) | 3 (3)
10016791-Flu like symptoms (General disorders) | 2 (2)
10017577-Gait disturbance (General disorders) | 3 (3)
10033371-Pain (General disorders) | 9 (9)
10050068-Edema limbs (General disorders) | 2 (2)
10062466-Localized edema (General disorders) | 1 (1)
10062501-Non-cardiac chest pain (General disorders) | 3 (3)
10040753-Sinusitis (Infections and infestations) | 1 (1)
10040872-Skin infection (Infections and infestations) | 2 (2)
10046300-Upper respiratory infection (Infections and infestations) | 3 (3)
10046571-Urinary tract infection (Infections and infestations) | 2 (2)
10061229-Lung infection (Infections and infestations) | 1 (1)
bacterial infection (Infections and infestations) | 1 (1)
10016173-Fall (Injury, poisoning and procedural complications) | 1 (1)
10001551-Alanine aminotransferase increased (Investigations) | 5 (5)
10001675-Alkaline phosphatase increased (Investigations) | 11 (11)
10003481-Aspartate aminotransferase increased (Investigations) | 10 (10)
10005364-Blood bilirubin increased (Investigations) | 5 (5)
10008661-Cholesterol high (Investigations) | 2 (2)
10011368-Creatinine increased (Investigations) | 16 (16)
10025256-Lymphocyte count decreased (Investigations) | 10 (10)
10029366-Neutrophil count decreased (Investigations) | 6 (6)
10035528-Platelet count decreased (Investigations) | 13 (13)
10047896-Weight gain (Investigations) | 5 (5)
10047900-Weight loss (Investigations) | 16 (16)
10049182-White blood cell decreased (Investigations) | 14 (14)
10055599-Hemoglobin increased (Investigations) | 2 (2)
10056910-GGT increased (Investigations) | 4 (4)
10002646-Anorexia (Metabolism and nutrition disorders) | 9 (9)
10012174-Dehydration (Metabolism and nutrition disorders) | 1 (1)
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 10 (10)
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
10020680-Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (5)
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (14)
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 15 (15)
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 10 (10)
10021018-Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
10021038-Hyponatremia (Metabolism and nutrition disorders) | 17 (17)
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
10029883-Obesity (Metabolism and nutrition disorders) | 1 (1)
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
10003246-Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10031282-Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
10048677-Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10048706-Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
10065895-Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion with extensive nodular synovial proliferation (Musculoskeletal and connective tissue disorders) | 1 (1)
urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
10013573-Dizziness (Nervous system disorders) | 6 (6)
10013911-Dysgeusia (Nervous system disorders) | 3 (3)
10019211-Headache (Nervous system disorders) | 6 (6)
10024264-Lethargy (Nervous system disorders) | 2 (2)
10033987-Paresthesia (Nervous system disorders) | 2 (2)
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
10041349-Somnolence (Nervous system disorders) | 3 (3)
10051272-Facial muscle weakness (Nervous system disorders) | 1 (1)
piriformis syndrome (Nervous system disorders) | 1 (1)
10002855-Anxiety (Psychiatric disorders) | 3 (3)
10022437-Insomnia (Psychiatric disorders) | 2 (2)
10019450-Hematuria (Renal and urinary disorders) | 1 (1)
10037032-Proteinuria (Renal and urinary disorders) | 6 (6)
10046539-Urinary frequency (Renal and urinary disorders) | 1 (1)
10046555-Urinary retention (Renal and urinary disorders) | 1 (1)
10046628-Urine discoloration (Renal and urinary disorders) | 1 (1)
10061574-Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
10062225-Urinary tract pain (Renal and urinary disorders) | 1 (1)
10034263-Pelvic pain (Reproductive system and breast disorders) | 2 (2)
10046904-Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
10046916-Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10036790-Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10047681-Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
10015218-Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
10040868-Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
10040947-Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
hand-foot syndrome symptoms (Skin and subcutaneous tissue disorders) | 1 (1)
10016825-Flushing (Vascular disorders) | 1 (1)
10020407-Hot flashes (Vascular disorders) | 2 (2)
10020772-Hypertension (Vascular disorders) | 25 (25)
10021097-Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01157091/Prot_SAP_000.pdf